CLINICAL TRIAL: NCT05903131
Title: UPLifT-Endo: Uterine Preservation Via Lifestyle Transformation A Behavioral Intervention to Promote Primary Prevention and Uterine Preservation in Premenopausal Women With Obesity and Atypical Endometrial Hyperplasia or Grade 1 Endometrial Cancer
Brief Title: Uterine Preservation Via Lifestyle Transformation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 202307204; P50CA265793 (NIH)
Record Dates: First submitted 2023-05-24; First posted 2023-06-15 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Hyperplasia; Grade 1 Endometrial Cancer
Keywords: fertility-sparing; weight management; obesity; endometrial cancer; behavioral intervention; premenopausal endometrial hyperplasia; premenopausal endometrial cancer
MeSH Terms: conditions — Endometrial Hyperplasia; Obesity; Endometrial Neoplasms | interventions — Progestins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Levonorgestrel-releasing IUD (LNG-IUD) + Behavioral Weight Loss Intervention (Experimental): * The levonorgestrel-releasing IUD is used in this study as per standard care.
  * The behavioral weight loss intervention consists of a telemedicine cognitive behavioral coaching program. At each session, patients will self-report weight, number of days they kept a food journal during the past week, average daily caloric intake for the week, number of days exercised for the week, total number of minutes of moderate physical activity, and average number of steps per day for the week.
  Interventions: Behavioral: Telemedicine behavioral weight intervention; Drug: Progestin; Drug: Levonorgestrel-releasing IUD.
- Arm 2: Levonorgestrel-releasing IUD (LNG-IUD) + Enhanced Usual Care (Active Comparator): * The levonorgestrel-releasing IUD is used in this study as per standard care.
  * Participants will be provided with 1- to 3-page handouts on topics including healthy eating, exercise, and behavioral eating strategies from materials provided on the American Cancer Society, Society of Gynecologic Oncology, and WebMD Nourish websites. These materials encourage weight loss through calorie counting, recording dietary intake, engaging in exercise programs, and using portion control strategies.
  * The participants randomized to this arm will cross over to the behavioral weight loss intervention arm at 12 months if they have not achieved resolution of AEH or grade 1 endometrial cancer.
  Interventions: Behavioral: Enhanced usual care; Drug: Levonorgestrel-releasing IUD.

INTERVENTIONS:
Behavioral: Telemedicine behavioral weight intervention — Weekly telephone calls during the first month, biweekly during the next 5 months, and then monthly for the last 7 months (12 months total). Each telephone session will be 30 minutes long.
  Arms: Arm 1: Levonorgestrel-releasing IUD (LNG-IUD) + Behavioral Weight Loss Intervention
Drug: Progestin — Released via the levonorgestrel-releasing IUD.
  Arms: Arm 1: Levonorgestrel-releasing IUD (LNG-IUD) + Behavioral Weight Loss Intervention
Behavioral: Enhanced usual care — 1-3 page handouts
  Arms: Arm 2: Levonorgestrel-releasing IUD (LNG-IUD) + Enhanced Usual Care
Drug: Levonorgestrel-releasing IUD. — Standard of care

SUMMARY:
Up to 60% of endometrial cancer cases are attributed to obesity, in part because obesity promotes development of atypical endometrial hyperplasia (AEH), and up to 40% of women with AEH go on to develop endometrial cancer. The increasing prevalence of obesity in premenopausal women has resulted in increasing rates of AEH in this age group. Hysterectomy with removal of the fallopian tubes and ovaries is 100% effective in preventing endometrial cancer, but this approach results in infertility. Fertility-sparing treatments exist, such as treatment with oral or intrauterine progestin, but these treatments do not work uniformly and do not combat the underlying cause of endometrial cancer, which is obesity and metabolic syndrome. Additionally, up to 41% of women on progestin eventually experience relapse of AEH or endometrial cancer. Third, many patients have insulin resistance that may worsen with progestin therapy. Thus, to improve treatment of AEH and grade 1 endometrial cancer, prevent and reverse endometrial cancer, and allow women to preserve their fertility, the investigators must integrate an effective weight loss strategy to be given with progestin treatment. It is the hypothesis that premenopausal women with AEH desire uterine preservation will be more likely to have atypia-free uterine preservation at one year if they receive progestin in combination with a behavioral weight loss intervention versus progestin plus enhanced usual care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histologically confirmed complex atypical endometrial hyperplasia (AEH) or grade 1 endometrial cancer.

  * Patients with a previous diagnosis of AEH or grade 1 endometrial cancer who are already being followed with conservative management with oral or LNG-IUD progestin therapy are eligible.
  * For patients with a previous diagnosis of AEH or grade 1 endometrial cancer who have been placed on progestin prior to study entry, the duration of IUD or oral progestin use prior to trial entry should be documented.
* Premenopausal woman with a uterus.
* ECOG performance status of 0-2.
* At least 18 years of age and no more than 45 years of age.
* Undergoing uterine-sparing management (e.g. due to interest in fertility preservation, interest in uterine preservation, provider recommendation, or other reason).
* BMI ≥ 30 kg/m^2.
* Prior or current receipt of progestin is allowed as above. Willingness to undergo placement of LNG-IUD at the time of study entry.
* Ability to understand and willingness to sign an IRB approved written informed consent document.

Exclusion Criteria:

* Current, active treatment for any malignant neoplasm with chemotherapy or radiation.
* Pregnant and/or breastfeeding. Participants must have a negative urine or serum pregnancy test during screening window and within 7 days prior to LNG-IUD insertion. If LNG-IUD is in place, lack of pregnancy is assumed.
* Active pelvic infection at the time of IUD placement or other contraindication to the use of an IUD in the opinion of the treating physician.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with atypical endometrial hyperplasia (AEH)-free biopsy | At 1 year

SECONDARY OUTCOMES:
Time to resolution of atypical endometrial hyperplasia (AEH) | Through completion of follow-up (estimated to be 2 years)
  Defined as the period of time in months/days from the first biopsy to show AEH or grade 1 endometrial cancer to the first biopsy that shows no evidence of hyperplasia or malignancy
Time to resolution of endometrial cancer | Through completion of follow-up (estimated to be 2 years)
Atypia-free survival | Through completion of follow-up (estimated to be 2 years)
  -Defined as the time interval from the date of positive treatment response (as determined by biopsy) to the date of atypical endometrial hyperplasia (AEH) recurrence. AEH-free or the patients with lost to follow-up will be censored at the last follow-up.
Endometrial cancer progression-free survival (EC-PFS) | Through completion of follow-up (estimated to be 2 years)
  EC-PFS is defined as the time interval from the date of positive treatment response (as determined by biopsy) to the date of recurrence of EC. Endometrial cancer-free patients or the patients with lost to follow-up will be censored at the last follow-up.
Change in weight | Through completion of follow-up (estimated to be 2 years)
Change in Cancer Worry Impact Events Scale (CWIES) | At enrollment, 6 months, 12 months, end of intervention, and 24 months (estimated to be 2 years)
  The CWIES is a 15-item self-report measure evaluating stress reactions and traumatic experiences, specifically inquiring about cancer worry-specific distress. Range of values for each individual item will be a Likert Scale from 0-5. 0=not at all and 5=often. The higher the score, the more cancer-worry specific distress the participant has.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea R Hagemann, M.D., MSCI, Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (3):
  - Washington University School of Medicine, St Louis, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - University of Oklahoma, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu